CLINICAL TRIAL: NCT06759259
Title: Mannitol Adjuvant Administration for Delerium Prevention
Brief Title: Mannitol Administration for Delerium Prevention
Acronym: MAD
Status: Completed | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 231
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Infarction (MI); Delirium, Intensive Care Unit, Randomised Controlled Trial
Keywords: myocardial infarction; delirium; prevention; inflammation
MeSH Terms: conditions — Myocardial Infarction; Delirium; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate the efficacy of adjuvant administration of mannitol for the prevention of delirium in patients with myocardial infarction.

DETAILED DESCRIPTION:
The pathogenesis of delirium in patients with myocardial infarction has not been fully studied, as a result of which delirium is currently considered a polyetiological syndrome. The ideas about the pathogenesis of delirium are formulated in a number of concepts, among which the neuroinflammatory theory is the most promising for study. The development of a systemic inflammatory reaction of both infectious and aseptic nature can lead to a violation of the permeability of the blood-brain barrier, followed by subclinical cerebral edema and impaired neurotransmitter metabolism. A single study of the adjuvant use of mannitol for the prevention of delirium, conducted in 2020 (Hamiko M.) proved the effectiveness of mannitol in the prevention of delirium in patients who underwent surgical aortic valve replacement, and served as a theoretical and experimental prerequisite for this study.

The study is prospective, randomized, open-label, controlled. It is planned to include 40 patients with myocardial infarction aged 65 years or older on the first day of the disease ("pain-door" < 24 hours) and signs of a systemic inflammatory response (CRP> 25 mg / L) in the main and control groups in a 1: 1 ratio. All patients will receive standard treatment for myocardial infarction upon admission in accordance with current recommendations. Patients will be randomized using a random number generator, after which patients in the main group will receive adjuvant therapy with mannitol at a dose of 1000 mg / kg according to the following scheme: bolus 250 mg / kg + infusion 66.6 mg / kg / hour until a total dose of 1000 mg / kg is reached. Patients in the control group will receive standard treatment for myocardial infarction. It is planned to evaluate clinical, laboratory, functional data and take blood samples for the study of markers of systemic inflammation and brain damage and other biomarkers on days 1, 3 and 7. Evaluation of remote outcomes is planned on days 30 and 90.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and over
* Myocardial infarction in the first day of illness ("pain to door" time < 254 hours)
* Serum CRP > 25 mg/L

Exclusion Criteria:

* A known pathological process in the brain, psychiatric disorders
* Impossibility of conducting an assessment CAM-ICU

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients in the first day of development of myocardial infarction with signs of systemic inflammation and initial normal mental status and the absence of previously known pathological processes of the brain and psychiatric disorders.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-12-29 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
delirium | 1-14 days
  Development of delirium during hospitalization

SECONDARY OUTCOMES:
In-hospital mortality | 1-30 days
  Death during hospitalization from all causes
In-hospital LOS | 1-30 lays
  Lenght of stay in hospital
ICU-LOS | 1-30 days
  Lenght of stay in ICU
Re-hospitalization due to MACE | 1-90 days
  Re-hospitalization due to MACE

OTHER OUTCOMES:
Dynamics of brain damage markers | 1, 3, 7 days
  Dynamics of brain damage markers (NSE, S100β)
Dynamics of markers of systemic inflammation | 1, 3, 7 days
  Dynamics of markers of systemic inflammation (IL-1, IL-6, IL-8, procalcitonin, presepsin)
Early adverse LV remodeling | 1, 3, 7 days
  Increase in ESV by 15% from the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Panteleev, MD, Principal Investigator — Tomsk NRMC
Locations (1):
- Cardiology Reserch Institute Tomsk National Research Centre, Tomsk, Tomsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: Undecided